CLINICAL TRIAL: NCT00946790
Title: Bioavailability of Hydroxychloroquine Sulfate, 200 mg Tablets
Brief Title: To Demonstrate the Relative Bioavailability of Hydroxychloroquine Sulfate, 200 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 005-14-10551
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Immunosuppression; Rheumatism
Keywords: Immunosuppressant and Antirheumatic
MeSH Terms: conditions — Rheumatic Diseases | interventions — Hydroxychloroquine; Trifyba

ARMS (2):
- 1 (Experimental): Hydroxychloroquine Sulfate Tablets, 200 mg (Geneva Pharmaceutical, Inc.)
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets, 200 mg (Geneva Pharmaceutical, Inc.)
- 2 (Active Comparator): Hydroxychloroquine Sulfate Tablets, 200 mg, Plaquenil (Sanofi Winthrop)
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets, 200 mg, Plaquenil (Sanofi Winthrop)

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets, 200 mg (Geneva Pharmaceutical, Inc.)
  Arms: 1
Drug: Hydroxychloroquine Sulfate Tablets, 200 mg, Plaquenil (Sanofi Winthrop)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of hydroxychloroquine sulfate, 200 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 1993-07; Primary Completion 1993-12 (Actual); Study Completion 1993-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 171 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gantt, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.